CLINICAL TRIAL: NCT01384045
Title: Randomized Trial of Health Promotion Outreach for Diabetes Cure
Brief Title: Outreach for Diabetes Cure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 08-0005
Record Dates: First submitted 2011-06-27; First posted 2011-06-28 (Estimated); Last update posted 2012-12-18 (Estimated); Status verified 2011-06

CONDITIONS: Type II Diabetes
Keywords: Type II Diabetes; Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual Care (No Intervention): Patients continue to receive usual diabetes care without outreach by health promotions staff.
- Arm 1-Health Promotoin Outreach (Experimental): Active outreach by health promotion staff to send diabetes report card and schedule services including laboratory testing and visits.
  Interventions: Other: Health promotion outreach

INTERVENTIONS:
Other: Health promotion outreach — Calling patients who are due for diabetes related services, sending them an interventional letter and assisting them in getting over due serves.
  Arms: Arm 1-Health Promotoin Outreach

SUMMARY:
Using a socioeconomic, race/ethnic, and gender-diverse sample of patients who receive diabetes care from a University of Colorado Hospital (UCH) primary care provider (PCP), carry out a randomized-controlled trial of usual care versus an outreach intervention designed to increase guideline concordance with American Diabetes Association (ADA) recommendations for blood pressure, Low-density lipoprotein (LDL), and glycosylated hemoglobin (A1c) goals, referrals for retinal exams, and aspirin therapy.Primary hypotheses: The proportion of patients meeting goal will be 10% higher in the intervention compared with control group in the following domains: 1. LDL<100 mg/dL; 2. A1c<7.0%; and 3. Systolic blood pressure<130 mm Hg or diastolic blood pressure<80 mm Hg.

DETAILED DESCRIPTION:
Ten percent of all people over the age of 20, and 21% of all people over the age of 60, have diabetes. Diabetes is the sixth leading cause of death, and is one of the most prominent causes of heart disease, stroke, blindness, nephropathy, and neuropathy. Total health care expenditures for diabetes and its complications are enormous, amounting to more than $132 billion in direct and indirect costs in 2002. Nationally, substantial percentages of diabetic patients are not meeting ADA, Health Plan Employer Data and Information Set, (HEDIS), and Physician Quality Reporting Initiative (PQRI) guidelines for care that are intended to reduce morbidity and mortality associated with this disease. In order to improve these statistics, novel ways of delivering primary and secondary preventive diabetes care are needed. The growing use of electronic medical record systems and the ability to extract clinically-relevant information from administrative data sets offer powerful opportunities to identify patients who are "falling through the cracks," reach out to them proactively where they live, and render medical services and education in ways that maximize convenience and minimize barriers associated with sporadic and time-limited clinic visits.

The delivery of preventive and chronic disease services is sub-optimal in outpatient settings. Rates of guideline concordance for diabetes care within University of Colorado Hospital (UCH) are in most instances modestly better than national averages, yet there remains tremendous room for improvement. Clinic visits are often too brief for medical providers to review and arrange for all recommended care. Providers are frequently hampered by poorly-organized clinical data and a lack of automated reminders. Finally, many patients do not know about recommendations for care and prefer to focus on acute concerns during clinic visits.

Although decision support in the medical provider's office can improve guideline-based care for chronic illness, it does not improve outcomes among patients who fail to make clinic appointments or who make appointments for reasons unrelated to the illness. The investigators developed a health promotion outreach system (HPOS) to overcome many of these barriers. The purpose of HPOS is to increase access to and enhance the delivery of guideline-based care by communicating with patients outside of clinical settings.

Our diabetes-specific HPOS intervention incorporates the following key elements: (1) electronic queries of administrative claims to identify patients who are not up-to-date with recommended diabetes services; (2) mail and telephone outreach to alert patients about recommendations for care and facilitate the direct scheduling of primary care provider (PCP) visits, laboratory testing several days before PCP visits, and ophthalmology appointments; and (3) advance PCP notification regarding the intended diabetes focus of appointments arranged through the outreach process. The purpose of this study is to assess whether this intervention improves guideline concordance for LDL cholesterol, hemoglobin A1c, blood pressure, retinal examinations, and aspirin therapy as well as clinical attention to diabetes during primary care visits.

The investigators believe our intervention will reduce several barriers associated with usual care. First, the investigators reach out proactively to inform patients about recommendations for care instead of waiting for them to make appointments haphazardly and often for reasons unrelated to diabetes. The investigators make daytime and evening telephone calls to patients, many of whom are undoubtedly busy and forgetful, when they do not themselves call in response to letters that summarize personalized recommendations. The investigators schedule all laboratories and PCP visits at a single point in time, over the phone, and then send reminder postcards that summarize this information. Rather than completing laboratory testing during PCP visits and then requiring PCPs to convey recommendations for care several days later, the investigators schedule laboratories ahead of time whenever possible so that timely information will be available help guide clinical decision-making at the point of care. Finally, the investigators notify patients and PCPs in advance about the diabetes-specific purpose of scheduled appointments and specific areas needing clinical attention.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of type II diabetes
* visit to University of Colorado Hospital in primary care clinic in last 18 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2800 (Actual)
Dates: Start 2009-02; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Composite Measure of Guideline Concordance | After 1 year
  Composite measure of guideline concordance with 1 point for concordance with each of the following:
  1. hemoglobin a1c less than 7%
  2. ldl cholesterol less than 100 mgs per decaliter
  3. urinary micro albumin measured in preceding 12 months
  4. both systolic bp less than 130 mms mercury & diastolic bp less than 80 mms mercury

SECONDARY OUTCOMES:
Individual measures of guideline concordance | After 1 year
  Individual measures of guideline concordance. Assessment of the outcome measures of the composite measures separately.

CONTACTS AND LOCATIONS:
Overall Officials: Steven Ross, MD, Principal Investigator — University of Colorado, Denver; Razzaghi Mitra, MD, Principal Investigator — University of Colorado, Denver; Lobo Ingrid, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Hopspital, Aurora, Colorado, United States